CLINICAL TRIAL: NCT01759433
Title: Reference Ranges for Sonoclot Analysis in Chinese
Brief Title: Reference Intervals for Sonoclot Analysis in Chinese
Status: Completed | Type: Observational
Sponsor: Wuhan Asia Heart Hospital (Other)
Responsible Party: Principal Investigator, Zhenlu Zhang, Director of the clinical laboratory, Wuhan Asia Heart Hospital
Other Study IDs: SCWH001
Record Dates: First submitted 2012-11-29; First posted 2013-01-03 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — 2.7 mL citrated blood.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The reference intervals for Sonoclot Analysis may be different between Chinese and American. So far, no reference interval has been established in Chinese for Sonoclot Analysis. This study is going to establish the first Chinese reference intervals for Sonoclot Analysis and test whether they are different from American reference intervals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Han ethnic

Exclusion Criteria:

* Renal dysfunction
* Liver disorders
* Known coagulation disorders
* Patients taking medications in the last month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese healthy adults aged 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The reference intervals for sonoclot analysis in Chinese | 3 month
  whether Chinese reference intervals are different from Caucasian reference intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Asia Heart hospital, Wuhan, Hubei, China